CLINICAL TRIAL: NCT00156117
Title: A Multicenter, Randomized, Double-Blind, Fixed-Dose, 6-Week Trial of the Efficacy and Safety of Asenapine Compared With Placebo Using Olanzapine Positive Control in Subjects With an Acute Exacerbation of Schizophrenia
Brief Title: Efficacy and Safety of Asenapine With Placebo and Olanzapine (41021)(P05933)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05933; Hera; 41021
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): asenapine 5 mg BID and 10 mg BID
  Interventions: Drug: asenapine
- 2 (Placebo Comparator): Placebo against olanzapine and asenapine
  Interventions: Drug: Placebo
- 3 (Active Comparator): olanzapine 15 mgQD
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: asenapine — 5 mg BID or 10mg BID
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2
Drug: olanzapine — olanzapine 15 mg QD
  Arms: 3

SUMMARY:
Schizophrenia is a brain disease. The primary features of schizophrenia are characterized by Positive symptoms (symptoms that should not be there, inability to think clearly, to distinguish reality from fantasy i.e., hearing voices) and Negative symptoms (a reduction or absence of normal behaviors or emotions, i.e., unable to manage emotions, make decisions and relate to others). Other symptoms include reduced ability to recall and learn new information, difficulty with problem solving, or maintaining productive employment. The symptoms of schizophrenia may be due to an imbalance in chemicals in the brain, primarily dopamine and serotonin, which enables brain cells to communicate with each other.

Asenapine is an investigational drug that may help to correct the imbalance in dopamine and serotonin. This is a 6 week study to test the efficacy and safety of asenapine and a comparator agent (olanzapine) in the treatment of patients with schizophrenia. Patients that complete this trial will have the option of continuing in an additional one year extension trial.

ELIGIBILITY:
Inclusion Criteria:

* Currently suffering from an acute exacerbation of schizophrenia. Caregiver required.

Exclusion Criteria:

* Have an uncontrolled, unstable medical condition. Have any other psychiatric disorder other than schizophrenia as a primary diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2005-05-12 (Actual); Primary Completion 2006-04-28 (Actual); Study Completion 2006-05-30 (Actual)

PRIMARY OUTCOMES:
Change in total PANSS score at endpoint (6-week double-blind or last assessment after baseline) from baseline | Screen, baseline, Days 4,7,14,21,28,35,42

SECONDARY OUTCOMES:
Changes in PANSS subscale and Marder factor scores; CGI-S scores | Screen, baseline, Days 4,7,14,21,28,35,42
CGI-I scores | Days 4,7,14,21,28,35,42
Neurocognition and cognitive functioning | Baseline , day 42
Anxiety | Baseline, day 42
Suicidal thinking | Baseline, day 42
Quality of life and patient functionality | Baseline, day 42
Readiness to discharge, at scheduled assessments and endpoint from baseline | Baseline up to day 14
Extrapyramidal symptoms | Baseline, Days 4,7,14,21,28,35,42
Laboratory parameters | Baseline, Days 14,,28,,42
Vital signs | Baseline, Days ,14,21,28,42
Weight | Baseline, Days 14,,28,,42
ECGs | Baseline, Days ,14,,28,,42
Adverse events (including serious adverse events) | Screen, baseline, Days 4,7,14,21,28,35,42 and are are recorded continuously for AEs up to 7 days after endpoint
SAEs up to 30 days after endpoint | Screen, baseline, Days 4,7,14,21,28,35,42 and are are recorded continuously for AEs up to 30 days after endpoint

REFERENCES:
- [Result] Szegedi A, Verweij P, van Duijnhoven W, Mackle M, Cazorla P, Fennema H. Meta-analyses of the efficacy of asenapine for acute schizophrenia: comparisons with placebo and other antipsychotics. J Clin Psychiatry. 2012 Dec;73(12):1533-40. doi: 10.4088/JCP.11r07596. PMID 23290326
- [Derived] Castle DJ, Slott Jensen JK. Management of depressive symptoms in schizophrenia. Clin Schizophr Relat Psychoses. 2015 Apr;9(1):13-20. PMID 25367164